CLINICAL TRIAL: NCT02664831
Title: Immunoinflammatory and Metabolic Responses in Post Cardiac Arrest Syndrome (PCAS)
Brief Title: Immunoinflammatory Response in Post Cardiac Arrest Syndrome (PCAS)
Acronym: PCAS
Status: Recruiting | Type: Observational
Sponsor: MaineHealth (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David B. Seder MD, Chair, Department of Critical Care Services, MaineHealth
Other Study IDs: DBS1; 1P20GM139745-01 (NIH)
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Arrest; Inflammation; Obesity; Hypoxic Ischemic Encephalopathy (HIE)
Keywords: cardiac arrest; inflammation; immune; neuregulin; lymphocyte; neutrophil; brown adipose; HIE
MeSH Terms: conditions — Heart Arrest; Inflammation; Obesity; Hypoxia-Ischemia, Brain; Fibromatosis, Gingival, 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Red blood cells and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective, observational study to investigate molecular mechanisms mediating the systemic inflammatory process, and changes to metabolism, and their impact on brain injury, survival, and functional outcomes after cardiac arrest. Investigators have shown that cardiac arrest induces changes in the numbers and properties of circulating immune cells, shifting the balance towards a pro-inflammatory phenotype and there is increased interest in the inflammatory pathways and the signaling mechanisms through which they are modulated. Participants will undergo blood sampling during 7 days following cardiac arrest, and analyses performed. Patient characteristics, clinical circumstances, and outcomes will be recorded and their associations with these inflammatory pathways characterized.

DETAILED DESCRIPTION:
Preliminary evidence indicates that inter-individual variables such as immune cell activity and the production of pro-inflammatory factors may differentiate patients with the highest risk of poor neurological outcome, and may reveal novel therapeutic approaches based on promoting molecular pathways of inflammation-resolution and recovery to reduce the severity of hypoxic ischemic encephalopathy (HIE). Additionally, there are intrinsic, modifiable metabolic factors, such as the presence and metabolic activity of brown adipose tissue (BAT) that may modulate injury and recovery.

Comparative analysis showed that cardiac arrest survivors have more CD73+ lymphocytes compared to non-survivors. CD73 is the key enzyme in the generation of anti-inflammatory and immunosuppressive adenosine. We have also identified novel populations of neutrophils (CD14posCD16low and DEspR+) that had amplified response to inflammatory stimuli. The investigators hypothesize that individual variability in the expression and signaling profiles of white blood cells (lymphocytes, neutrophils, monocytes and macrophages) following resuscitation affects inflammation and is independently associated with neurological outcome. To test this hypothesis, investigators will determine levels of various immune cell populations at different time points in peripheral blood of patients. Characterization of blood circulating factors, clinical phenotypes, and neurological outcomes after cardiac arrest is a second aim of this project, with a focus on understanding the heterogeneity of cellular and humoral immune responses and how they relate to different clinical phenotypes of post-resuscitation syndrome.

PCAS metabolism:

IT is known that hyperglycemia is an independent risk factor for poor outcome after cardiac arrest, but it is not known if modification of hyperglycemia reduces this risk. Published studies have not demonstrated benefit with intensive insulin therapy. Our preliminary data suggest correlation between brown adipose tissue activity and good outcome. We have postulated that BAT may be activated by therapeutic hypothermia and may act as a glucose sink reducing the oxidative stress caused by hyperglycemia, and secondarily reducing injury to the brain, heart, and other organs.

In these studies we will also investigate other actionable targets for new therapies.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Admitted to the intensive care unit after cardiac arrest episode
* Unresponsive after resuscitation

Exclusion Criteria:

* Moribund / actively dying at the time of evaluation
* Informed consent cannot be obtained within 24 hours of resuscitation
* Hemoglobin less than 7.0 g/dL, active high-volume bleeding, or requiring a transfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiac arrest survivors with encephalopathy admitted to the intensive care unit and unresponsive after resuscitation
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Correlations between inflammatory markers and clinical outcomes | 14 days
  Correlations between inflammatory markers and clinical outcomes
Correlations between inflammatory markers and biomarkers of neurological and cardiac injury | 7 days
  Correlations between inflammatory markers and biomarkers of neurological and cardiac injury

SECONDARY OUTCOMES:
Characterization of post-resuscitation inflammatory mechanisms and their regulators | 7 days
  Characterization of post-resuscitation inflammatory mechanisms and their regulators
Brown Fat activity | 2 weeks
  Correlations between 12,13 diHOME, blood glucose, and outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Ryzhov, MD, PhD, Principal Investigator — MaineHealth Institute for Research; David B Seder, MD, Principal Investigator — MaineHealth
Locations (1):
- Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in any publications, after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 6 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee.
URL: https://www.mainehealth.org/providers/david-b-seder-md

REFERENCES:
- [Background] deKay JT, Chepurko E, Chepurko V, Knudsen L, Lord C, Searight M, Tsibulnikov S, Robich MP, Sawyer DB, Gagnon DJ, May T, Riker R, Seder DB, Ryzhov S. Delayed CCL23 response is associated with poor outcomes after cardiac arrest. Cytokine. 2024 Apr;176:156536. doi: 10.1016/j.cyto.2024.156536. Epub 2024 Feb 6. PMID 38325139
- [Background] Ryzhov S, May T, Dziodzio J, Emery IF, Lucas FL, Leclerc A, McCrum B, Lord C, Eldridge A, Robich MP, Ichinose F, Sawyer DB, Riker R, Seder DB. Number of Circulating CD 73-Expressing Lymphocytes Correlates With Survival After Cardiac Arrest. J Am Heart Assoc. 2019 Jul 2;8(13):e010874. doi: 10.1161/JAHA.118.010874. Epub 2019 Jun 25. PMID 31237169